CLINICAL TRIAL: NCT03850002
Title: Lung Clearance Index for the Early Detection and Monitoring of Lung Allograft Dysfunction After Adult Lung Transplantation
Brief Title: Lung Clearance Index and Lung Allograft Dysfunction
Status: Withdrawn | Type: Observational
Why Stopped: PI leaving institution
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-02174
Record Dates: First submitted 2019-02-14; First posted 2019-02-21 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Lung Transplantation; Chronic Lung Allograft Dysfunction; Rejection Lung Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Early detection of CLAD by Lung Clearance Index (LCI) — Lung transplant candidates without prior CLAD (evaluated in study part I) will be followed over a period of 3 years to evaluate the potential of LCI to detect early CLAD

SUMMARY:
The aim of this project is to evaluate the ability of the lung clearance index (LCI) to detect early chronic lung allograft failure (CLAD) in adult lung transplant recipients over a period of 3 years.

DETAILED DESCRIPTION:
This single center study consists of three parts:

1. Characterisation of the Zurich lung transplant cohort regarding CLAD status and pulmonary function impairment (cross-sectional, study part I)
2. Evaluation of test-retest reliability of LCI in 20 clinically stable lung transplant recipients during three consecutive study visits (study part II)
3. Prospective cohort study to test the ability of LCI to detect early CLAD in patients without prior CLAD (study part III)

ELIGIBILITY:
Inclusion Criteria:

* Male and female lung transplant recipients
* Written informed consent by the participant after information about the research project

Exclusion Criteria:

* Any contraindication to perform pulmonary function tests (e.g., persistent pneumothorax)
* Acute airway infection
* Chronic infection due to Burkholderia spp and nontuberculosis mykobacteria NTM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult lung transplant patients from University Hospital Zurich will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in lung clearance index (LCI) | Change from baseline up to 3 years
  Measured by multiple breath nitrogen washout (Exhalyzer® D; Eco Medics AG)

SECONDARY OUTCOMES:
Change in slope of acinar airways (Sacin) | Change from baseline up to 3 years
  Measured by multiple breath nitrogen washout (Exhalyzer® D; Eco Medics AG)
Change in slope of conducting airways (Scond) | Change from baseline up to 3 years
  Measured by multiple breath nitrogen washout (Exhalyzer® D; Eco Medics AG)
Change in forced expiratory volume in 1s (FEV1) | Change from baseline up to 3 years
  Measured by Spirometry (Geratherm Respiratory GmbH)
Change in forced vital capacity (FVC) | Change from baseline up to 3 years
  Measured by Spirometry (Geratherm Respiratory GmbH)
Change in forced expiratory flows at 25-75 of vital capacity (FEF25-75) | Change from baseline up to 3 years
  Measured by Spirometry (Geratherm Respiratory GmbH)
Change in total lung capacity (TLC) | Change from baseline up to 3 years
  Measured by Bodyplethysmography (Geratherm Respiratory GmbH)
Change in residual volume (RV) | Change from baseline up to 3 years
  Measured by Bodyplethysmography (Geratherm Respiratory GmbH)
Change in total lung capacity (TLC) / residual volume (RV) ratio | Change from baseline up to 3 years
  Measured by Bodyplethysmography (Geratherm Respiratory GmbH)
Change in diffusing capacity for nitric oxide (DLNO) | Change from baseline up to 3 years
  Single-breath measurements (Jaeger MasterScreenTM PFT system)
Change in diffusing capacity for carbon monoxide oxide (DLCO) | Change from baseline up to 3 years
  Single-breath measurements (Jaeger MasterScreenTM PFT system)
Change in DLNO/DLCO ratio | Change from baseline up to 3 years
  Single-breath measurements (Jaeger MasterScreenTM PFT system)
Change in transfer coefficient for nitric oxide (DLNO/VA) | Change from baseline up to 3 years
  Single-breath measurements (Jaeger MasterScreenTM PFT system)
Change in transfer coefficient for carbon monoxide (DLCO/VA) | Change from baseline up to 3 years
  Single-breath measurements (Jaeger MasterScreenTM PFT system)
Change in computed tomography score | Change from baseline up to 3 years
  Measured by Computed Tomography: Semiquantative score (i.e., Brody Score); Subscores including bronchiectasis, mucus plugging, airway wall thickening, consolidation, mosaic pattern and air trapping). Subscores will be expressed as the percentage of the maximum score on a scale of 0 (no disease) to 100 (maximal lung disease).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Benden, Prof., MD, Principal Investigator — University Hospital of Zurich, Zurich, Switzerland